CLINICAL TRIAL: NCT01609868
Title: The Effect of a Liquid Protein Modular on Growth and Outcomes in the NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Alegent Health Bergan Mercy Medical Center (Unknown)
Responsible Party: Principal Investigator, Corrine K. Hanson, PhD, IRB Administrator, University of Nebraska
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-16432
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Problem With Growth of an Infant
Keywords: premature infant feeding protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): infants in this arm will receive the current treatment that is standard of care for these infants, powder protein modular to achieve 4 gm/kg/day
  Interventions: Dietary Supplement: Powder protein modular
- experimental (Experimental): this group will receive a liquid protein modular that recently became commercially avaliable, to achieve the same protein of 4 grm/kg/day as the powder comparision group
  Interventions: Dietary Supplement: Liquid protein modular

INTERVENTIONS:
Dietary Supplement: Powder protein modular — Infants will receive powder protein modular to achieve 4 grm/kg/day
  Arms: control
Dietary Supplement: Liquid protein modular — Infants will receive a commerically avaliable liquid protein modular to provide 4 grm/kg/day
  Arms: experimental

SUMMARY:
The investigators hypothesis that premature infants receiving a commercially available liquid protein modular will have improved growth when compared with premature infants receiving a commercially available powder protein modular.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than 2000 gms at birth, receiving maternal breast milk

Exclusion Criteria:

* Infants receiving formula

Max Age: 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Growth in premature infants (percentile ranking at 36 weeks CGA) | birth to 36 weeks

SECONDARY OUTCOMES:
GI tolerance | birth to 36 weeks
  abdominal distention, feeding tolerance

CONTACTS AND LOCATIONS:
Locations (1):
- Alegent Bergan Hospital, Omaha, Nebraska, United States